CLINICAL TRIAL: NCT00570024
Title: The Effects of Traditional Acupuncture on Mechanisms of Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB# 7320; 1R01AT001482 (NIH)
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: Acupuncture; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TA (Active Comparator): Active TA
  Interventions: Procedure: Traditional Acupuncture
- AA (Other)
  Interventions: Procedure: AA
- Waiting Group (No Intervention)

INTERVENTIONS:
Procedure: Traditional Acupuncture — In Traditional acupuncture (TA), in which eight acupuncture points are selected, subjects will undergo three 30-minute sessions weekly for 12 weeks. Disposable acupuncture needles (1-1.5 inch sterilized stainless steel)will be inserted up to one inch deep through a plastic needle tube that is secured with adhesive tape to the skin.
  Arms: TA
Procedure: AA — In Traditional acupuncture (TA), in which eight acupuncture points are selected, subjects will undergo three 30-minute sessions weekly for 12 weeks. Disposable acupuncture needles (1-1.5 inch sterilized stainless steel)will be inserted up to one inch deep through a plastic needle tube that is secured with adhesive tape to the skin.
  Other Names: Alternative Acupuncture
  Arms: AA

SUMMARY:
This research is being done because sudden and unexpected cardiac death remains a significant problem in patients with established coronary heart disease and accounts for 30% of deaths in this group (150,000 deaths annually) despite recognition and treatment of their heart disease. A large body of evidence implicates psychosocial stress as a risk factor and trigger for reduced blood flow in the heart, heart attack and sudden cardiac death, yet the specific mechanisms of this relationship remain under investigation. The nervous system, which plays a role in regulation of the heart, can influence cardiac arrhythmias (irregular heart beats). There are several studies that suggest that acupuncture improves anginal symptoms (like chest pain or tightness) and blood pressure, while reducing stress and improving overall quality of life. The reason that acupuncture seems to have a positive effect on these factors is thought to be that it helps the arteries and the nervous system to work better.

It is possible to measure these effects in a systematic way. The functioning of the artery can be measured by Peripheral Arterial Tonometry, (PAT) a simple monitoring device that measures blood flow using finger probes and a blood pressure cuff. Changes in the nervous system can be measured by using a 24-hour Holter monitor to record the heart rate. The 24-hour Holter monitor will also show if oxygen flow to the heart is decreased, as would happen during stress, by recording a continuous electrocardiogram (ECG). Feelings about stress can be established by questionnaires.

The purpose of this study is to compare three groups of people with known coronary heart disease. One group will receive traditional acupuncture, one group will receive alternative acupuncture, and a third group will receive usual care only.

DETAILED DESCRIPTION:
A. SPECIFIC AIMS Sudden and unexpected cardiac death remains a significant problem in patients with established coronary heart disease (CHD), and accounts for 30% of deaths in this group (~150,000 deaths annually) despite recognition and treatment of their disease. These sudden deaths are due to myocardial infarction and ischemic or nonischemically mediated arrythmias. Traditional risk factors do not completely account for the excess of CHD deaths. Although treatment of cardiac risk factors, such as hyperlipidemia, has been shown to significantly reduce cardiac events in populations with established coronary heart disease (e.g. by 34% in the Scandinavian Simvastatin Survival Study1) a majority of patients continue to have sudden and unexpected cardiac events including sudden cardiac death. Indeed, up to 50% of patients with established CHD will have recurrent events despite aggressive management of traditional risk factors such as hyperlipidemia, tobacco use and hypertension. This suggests that additional risk factors or mechanisms participate in the pathophysiological cascade underlying acute CHD events.

A large body of evidence implicates psychosocial stress as a risk factor and trigger for myocardial ischemia, infarction and sudden cardiac death, yet the specific mechanisms(s) of this relationship remain under investigation.2-9 The mechanisms may include hemodynamic, hemostatic and neuronally mediated effects on the cardiovascular system. Specifically they may include a prominent role of the cardiac autonomic nervous system, including the sympathetic nervous system (SNS) and parasympathetic nervous system (PNS).10 Indeed, cardiac arrhythmias have been implicated both as a risk factor and an etiology for sudden cardiac death, suggesting that alteration of cardiac autonomic nervous system tone may provide an opportunity for reducing acute cardiac events and sudden cardiac death. Prior work by ourselves and others has also demonstrated that sympathetic activation from psychosocial stress results in vascular constriction that, in the presence of impaired nitric oxide (NO) production and endothelial dysfunction, contributes to myocardial ischemia and adverse cardiac events, including sudden death. 6,8,11-15 Traditional Acupuncture (TA) is a Complementary and Alternative Medicine (CAM) practice with documented effects of improving physiologic imbalances and reducing psychosocial stress. For example, the TA technique has been shown, to significantly reduce mental stress in humans16, hypertension in an animal model17 and angina pectoris in CHD patients.18 These changes are consistent with the hypothesis that the TA technique directly alters autonomic nervous system tone, likely by reducing SNS activity, and possibly also by increasing PNS activity. We also hypothesize that TA may beneficially alter CHD indirectly by reducing psychosocial stress. Either of these hypotheses suggests that this CAM practice may serve as a complement or alternative to medical treatment for the prevention of acute cardiac events and sudden cardiac death.

We propose to evaluate the effect of TA on arterial vasomotor function and autonomic nervous system tone, two physiologic variables involved in the pathophysiological cascade underlying acute cardiac events and sudden death in CHD patients. To test for both the hypothesized direct and indirect effects of this CAM modality, we propose to compare an active TA intervention to two control groups: 1) an Alternative Acupuncture control group, and 2) a waiting control group, in patients with CHD.

Primary Aim

1. To assess effects of the TA technique (compared to Alternative Acupuncture and waiting control) on cardiac autonomic nervous system tone, as measured by heart rate variability (HRV) using Holter monitoring.

   Secondary Aims
2. To assess effects of the TA technique (compared to Alternative Acupuncture and waiting control) on CHD variables including a marker of inflammation (high sensitivity C reactive protein), symptoms (Seattle Angina Questionnaire), functional status (Duke Activity Status Inventory), blood lipoproteins, and blood pressure.
3. To assess effects of the TA technique (compared to Alternative Acupuncture and waiting control) on measures of perceived psychological stress, depression, hostility, anxiety, social support, and quality of life.

   Exploratory Aims
4. To estimate effect size of the TA technique (compared to Alternative Acupuncture and waiting control) on arterial vasomotor dysfunction, as measured by mental stress-brachial artery reactivity testing (BART) using high frequency ultrasound.

The results of the study will: a) provide an improved understanding of the hypothesized beneficial physiological and psychological effects of this CAM practice, and b) serve as potential pilot data for a multi-center TA proposal to evaluate the impact of TA on acute cardiac events, including sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Male or female
* Local residence
* Medically able to participate
* CAD by MI, CABG, PTCA, or stroke (>3 months prior), or angiographic evidence >50% epicardial coronary artery stenosis in at least one coronary artery
* Consent and referring MD approval

Exclusion Criteria:

* Comorbid disease precluding survival during study
* MI, unstable angina, CABG, PTCA or stroke within 3 months*
* HIV infection, chronic or active hepatitis or other blood-borne illness
* Cognitive, psychological or substance abuse-related impairment, as clinically assessed
* Atrial fibrillation, predominant pacemaker rhythm, significant conduction system disease, or automatic internal defibrillator*
* Significant valvular heart disease*
* Class III or IV heart failure*
* Renal or liver failure, as clinically assessed
* Participating in TA, or formal psychosocial stress management program
* Participation in another trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | 24 hours
  Holter monitoring will be recorded during the provocative procedures and during a 24-hour period during which subjects will document their activities and any anginal symptoms in a diary.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Bairey-Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

REFERENCES:
- [Background] Bots ML, Westerink J, Rabelink TJ, de Koning EJ. Assessment of flow-mediated vasodilatation (FMD) of the brachial artery: effects of technical aspects of the FMD measurement on the FMD response. Eur Heart J. 2005 Feb;26(4):363-8. doi: 10.1093/eurheartj/ehi017. Epub 2004 Dec 1. PMID 15618057
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Bonetti PO, Barsness GW, Keelan PC, Schnell TI, Pumper GM, Kuvin JT, Schnall RP, Holmes DR, Higano ST, Lerman A. Enhanced external counterpulsation improves endothelial function in patients with symptomatic coronary artery disease. J Am Coll Cardiol. 2003 May 21;41(10):1761-8. doi: 10.1016/s0735-1097(03)00329-2. PMID 12767662
- [Background] Chouraqui P, Schnall RP, Dvir I, Rozanski A, Qureshi E, Arditti A, Saef J, Feigin PD, Sheffy J. Assessment of peripheral artery tonometry in the detection of treadmill exercise-induced myocardial ischemia. J Am Coll Cardiol. 2002 Dec 18;40(12):2195-200. doi: 10.1016/s0735-1097(02)02591-3. PMID 12505234
- [Background] Goor DA, Sheffy J, Schnall RP, Arditti A, Caspi A, Bragdon EE, Sheps DS. Peripheral arterial tonometry: a diagnostic method for detection of myocardial ischemia induced during mental stress tests: a pilot study. Clin Cardiol. 2004 Mar;27(3):137-41. doi: 10.1002/clc.4960270307. PMID 15049379
- [Background] Moens AL, Goovaerts I, Claeys MJ, Vrints CJ. Flow-mediated vasodilation: a diagnostic instrument, or an experimental tool? Chest. 2005 Jun;127(6):2254-63. doi: 10.1378/chest.127.6.2254. PMID 15947345
- [Background] von Mering GO, Arant CB, Wessel TR, McGorray SP, Bairey Merz CN, Sharaf BL, Smith KM, Olson MB, Johnson BD, Sopko G, Handberg E, Pepine CJ, Kerensky RA; National Heart, Lung, and Blood Institute. Abnormal coronary vasomotion as a prognostic indicator of cardiovascular events in women: results from the National Heart, Lung, and Blood Institute-Sponsored Women's Ischemia Syndrome Evaluation (WISE). Circulation. 2004 Feb 17;109(6):722-5. doi: 10.1161/01.CIR.0000115525.92645.16. PMID 14970106
- [Derived] Mehta PK, Polk DM, Zhang X, Li N, Painovich J, Kothawade K, Kirschner J, Qiao Y, Ma X, Chen YD, Brantman A, Shufelt C, Minissian M, Merz CN. A randomized controlled trial of acupuncture in stable ischemic heart disease patients. Int J Cardiol. 2014 Sep 20;176(2):367-74. doi: 10.1016/j.ijcard.2014.07.011. Epub 2014 Jul 11. PMID 25103909